CLINICAL TRIAL: NCT03612531
Title: Manual Therapy for Fibrosis-Related Late Effect Dysphagia in Head and Neck Cancer Survivors: The Pilot MANTLE Trial
Brief Title: Manual Therapy in Treating Fibrosis-Related Late Effect Dysphagia in Head and Neck Cancer Survivors
Acronym: MANTLE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0052; NCI-2018-01511 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0052 (Other: M D Anderson Cancer Center); R21CA226200 (NIH)
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Cancer Survivor; Dysphagia; Fibrosis; Head and Neck Carcinoma
MeSH Terms: conditions — Deglutition Disorders; Fibrosis | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (manual therapy) (Experimental): Participants receive 10 manual therapy sessions performed by a speech pathologist during weeks 1-6. After completion of 6 weeks of therapy, participants perform manual therapy at home daily for 6 weeks.
  Interventions: Procedure: Manual Therapy

INTERVENTIONS:
Procedure: Manual Therapy — Receive manual therapy
  Other Names: MT

SUMMARY:
This trial studies how well manual therapy works in treating fibrosis-related late effect dysphagia in head and neck cancer survivors. Manual therapy is the use of massage and stretching exercises to increase blood flow and muscle movement in the neck, throat, jaw, and mouth, which may help to improve swallowing ability and range of motion in participants who have had treatment for head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and safety of manual therapy for treatment of fibrosis-related dysphagia in head and neck cancer survivors.

SECONDARY OBJECTIVES:

I.To estimate effect size, dose-response (number of treatment sessions to normalized cervical range of motion), and durability of manual therapy for improving cervical range of motion in head and neck cancer survivors with fibrosis-related late dysphagia.

II. To examine functional outcomes after manual therapy in head and neck cancer survivors with fibrosis-related late effects and their association with change in dysphagia grade, cervical extension, and other cofactors.

OUTLINE:

Participants receive 10 manual therapy sessions performed by a speech pathologist during weeks 1-6. After completion of 6 weeks of therapy, participants perform manual therapy at home daily for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Late Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) grade >= 2 dysphagia on Modified Barium Swallow (MBS) >= 2 years after curative-intent radiotherapy for head and neck cancer
* Grade >= 2 Common Terminology Criteria for Adverse Events (CTCAE) fibrosis
* Willing and able to return for 10 sessions over 6 weeks of therapy

Exclusion Criteria:

* Active recurrent or second primary head and neck, central nervous system, or thoracic cancer at time of enrollment
* Active osteoradionecrosis or other non-healing wounds (e.g., fistula, ulcer, soft tissue necrosis) in manual therapy (MT) regions of interest at time of enrollment
* History of subtotal or total glossectomy or total laryngectomy
* Functionally limiting cardiac, pulmonary, or neuromuscular disease
* Current tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Up to 12 weeks
  Will be determined by completion rate. Completion rate will be defined by completion of the 6 week clinical manual therapy (MT) program without withdrawing and attending a minimum of 2 sessions and the post-treatment assessment. Session attendance will be monitored separately to assess adherence and fidelity. Will summarize fidelity and adherence to the standard MT protocol using quantitative and qualitative methods.
Incidence of adverse events | Up to 12 weeks
  Will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Adverse events will be tabulated and will be monitored by the trial Data Safety Monitoring Board.

SECONDARY OUTCOMES:
Efficacy and durability of response | Up to 12 weeks; baseline, after manual therapy (6 weeks), and after home program wash-out period (6 weeks)
  Will be determined by cervical range of motion (CROM). CROM for each anatomic plane measured by goniometer.
Swallowing function and physiology | Baseline to 6 weeks (after manual therapy)
  Measured by videofluoroscopy using the Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) and Computational Analysis of Swallowing Mechanics (CASM).
Lingual and jaw range of motion (ROM) | Up to 12 weeks
  Measured by Therabite ruler.
Swallowing-related quality of life | Up to 12 weeks
  Measured by the MD Anderson Dysphagia Inventory (MDADI).
Symptom burden | Up to 12 weeks
  Measured by the MD Anderson Symptom Inventory Head and Neck Cancer Module (MDASI-HN).
Lymphedema/fibrosis staging | Up to 12 weeks
  Measured by the Common Terminology Criteria for Adverse Events and Head and Neck Lymphedema and Fibrosis Scale.
Performance status | Up to 12 weeks
  Measured by the Performance Status Scale for Head and Neck Cancer Patients (PSS-HN).
Soft tissue fibrosis | Up to 12 weeks
  Measured by magnetic resonance imaging.
Improvement in tongue innervation on Electromyography (EMG) findings | Baseline to 6 weeks (after manual therapy)
  Electromyography (EMG) scores are based on a 4-point denervation potentials grade with '0' being 'none' and '4' being 'full interference patterns of potentials'

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Hutcheson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] McMillan H, Warneke CL, Buoy S, Porsche C, Savage K, Lai SY, Fuller CD, Hutcheson KA. Manual Therapy for Fibrosis-Related Late Effect Dysphagia in Head and Neck Cancer Survivors: The MANTLE Nonrandomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2025 Apr 1;151(4):319-327. doi: 10.1001/jamaoto.2024.5157. PMID 39913160
- [Derived] Hutcheson K, McMillan H, Warneke C, Porsche C, Savage K, Buoy S, Wang J, Woodman K, Lai S, Fuller C. Manual Therapy for Fibrosis-Related Late Effect Dysphagia in head and neck cancer survivors: the pilot MANTLE trial. BMJ Open. 2021 Aug 4;11(8):e047830. doi: 10.1136/bmjopen-2020-047830. PMID 34348950
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org